CLINICAL TRIAL: NCT00989235
Title: A Phase 3B, Multi-Center, Randomized, Double-blind Study to Evaluate Remission and Joint Damage Progression in Methotrexate-naïve Early Erosive Rheumatoid Arthritis Subjects Treated With Abatacept Plus Methotrexate Compared With Methotrexate - Low Dose Sub-Study
Brief Title: Substudy - Low Dose of Abatacept in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-023 LT (Sub study); Eudrac # 2002-000784-26
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
Keywords: NOS
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abatacept (10 mg/Kg) (Active Comparator)
  Interventions: Drug: Abatacept
- Abatacept (5 mg/Kg) (Active Comparator)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — IV solution, IV, 10 mg/Kg, Once monthly, 1 year
  Other Names: BMS-188667
  Arms: Abatacept (10 mg/Kg)
Drug: Abatacept — IV solution, IV, 5 mg/Kg, Once monthly, 1 year
  Other Names: BMS-188667
  Arms: Abatacept (5 mg/Kg)

SUMMARY:
The purpose of this exploratory sub-study was to evaluate from a clinical perspective the impact on disease activity of lowering the dose of abatacept from 10 mg/kg to 5 mg/kg in subjects who had achieved remission (Disease Activity Score 28 [DAS 28]-erythrocyte sedimentation rate [ESR] < 2.6) at Day 701 of study IM101023.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the main study, are willing to participate and have a DAS 28 ESR score of < 2.6 on Day 701 of the main study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Westhovens R, Robles M, Ximenes AC, Wollenhaupt J, Durez P, Gomez-Reino J, Grassi W, Haraoui B, Shergy W, Park SH, Genant H, Peterfy C, Becker JC, Murthy B. Maintenance of remission following 2 years of standard treatment then dose reduction with abatacept in patients with early rheumatoid arthritis and poor prognosis. Ann Rheum Dis. 2015 Mar;74(3):564-8. doi: 10.1136/annrheumdis-2014-206149. Epub 2014 Dec 30. PMID 25550337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IM101023 (NCT00122382) was a 2-year study completing on Day 729, in which subjects were randomized to receive abatacept or placebo in combination with methotrexate (MTX) for the 1st year of the study and were then switched to open-label abatacept+MTX in the 2nd year. All subjects had received abatacept for a least 1 year prior start of sub-study.
Pre-assignment Details: Of the 433 participants who completed the main study (IM101-023 NCT00122382), 108 enrolled in the sub-study.
Groups:
- Abatacept (10 mg/kg): All subjects in the sub-study randomized to receive double-blind abatacept 10 mg/kg. Subjects rescued to open-label treatment received abatacept 10 mg/kg. The length of the sub-study is 1 year. As such, the maximum time the subject is treated collectively in double-blind and open-label treatment is 1 year.
- Abatacept (5 mg/kg): All subjects in the sub-study randomized to receive double-blind abatacept 5 mg/kg. Subjects rescued to open-label treatment received abatacept 10 mg/kg. The length of the sub-study is 1 year. As such, the maximum time the subject is treated collectively in double-blind and open-label treatment is 1 year.
Period: Overall Study
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Started | 58 | 50
Number Rescued to Open-Label Treatment | 4 | 4 (Of these, 1 was discontinued from open-label treatment (lost to follow-up).)
Number Completing Double-Blind Treatment | 51 | 41
Completed | 55 | 44
Not Completed | 3 | 6
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal of Consent | 1 | 1
Not completed — Desire to Become Pregnant | 1 | 0
Not completed — Randomized by Mistake | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Abatacept (10 mg/kg): All participants in the sub-study randomized to receive double-blind abatacept 10 mg/kg
- Abatacept (5 mg/kg): All participants in the sub-study randomized to receive double-blind abatacept 5 mg/kg
- Total: Total of all reporting groups
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg) | Total
Number analyzed (Participants) | 58 | 50 | 108
Age Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.5) | 51.1 (13.4) | 50.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 14 | 9 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Unknown | 2 | 0 | 2
  White | 49 | 46 | 95
  Black | 2 | 0 | 2
  Asian | 2 | 2 | 4
  Other | 3 | 2 | 5
Weight [Mean (Standard Deviation); unit: kg] — One participant in the 10 mg/kg group did not have weight reported.
  kg | 72.9 (14.7) | 73.8 (16.0) | 73.4 (15.3)
Disease Activity Scores Using C-reactive Protein (DAS 28 [CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 provides a score on a scale from 0 to 10 indicating the current activity of the rheumatoid arthritis (>5.1=high disease activity; <3.2=low disease activity; <2.6=remission).DAS 28 is a continuous variable which is a composite of 4 variables: the number of tender joints out of 28, the number of swollen joints out of 28 joints, C-reactive protein in mg/L (CRP) and subject assessment of disease activity measure on a visual analogue scale (VAS) of 100 mm based on the following formula:
  DAS 28 = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96.
  units on a scale | 2.1 (0.6) | 2.1 (0.6) | 2.1 (0.6)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Experiencing Disease Relapse
Description: Disease relapse is defined as additional DMARD therapy given, or 2 or more courses of high steroids given, or return to abatacept 10 mg/kg (rescue medication given), or DAS28 CRP score >= 3.2 at 2 consecutive visits.
Time Frame: After 12 Months of treatment
Population: Number of participants analyzed=number randomized.
Measure: Number; unit: Participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
Participants | 18 | 17

2. Secondary Outcome: Mean Time-Matched Baseline DAS28 CRP Scores
Description: Mean baseline DAS28 CRP values for the cohort of participants with serum samples available at that timepoint. DAS 28 is a continuous variable which is a composite of 4 variables: number of tender joints out of 28, number of swollen joints out of 28 joints, CRP in mg/L and subject assessment of disease activity measure on a visual analogue scale (VAS) of 100 mm. The DAS28 provides a score on a scale from 0 to 10 indicating the current activity of the rheumatoid arthritis (>5.1=high disease activity; <3.2=low disease activity; <2.6=remission).
Time Frame: Baseline
Population: Number of participants analyzed=number of participants randomized; n=All treated participants with available DAS28 CRP scores at that time point. Mean time-matched baseline values reflect changing n-values over time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
units on a scale
  Day 29 Cohort (n=45, 40) | 2.09 (0.61) | 2.05 (0.60)
  Day 57 Cohort (n=47, 37) | 2.06 (0.59) | 2.06 (0.62)
  Day 85 Cohort (n=46, 42) | 2.10 (0.60) | 2.09 (0.60)
  Day 113 Cohort (n=49, 39) | 2.06 (0.61) | 2.09 (0.62)
  Day 141 Cohort (n=47, 40) | 2.09 (0.59) | 2.10 (0.62)
  Day 169 Cohort (n=46, 36) | 2.10 (0.59) | 2.04 (0.61)
  Day 197 Cohort (n=44, 38) | 2.08 (0.60) | 2.06 (0.61)
  Day 225 Cohort (n=44, 38) | 2.09 (0.60) | 2.08 (0.63)
  Day 253 Cohort (n=46, 37) | 2.07 (0.60) | 2.04 (0.61)
  Day 281 Cohort (n=45, 38) | 2.07 (0.61) | 2.06 (0.61)
  Day 309 Cohort (n=45, 37) | 2.10 (0.58) | 2.08 (0.61)
  Day 337 Cohort (n=44, 36) | 2.09 (0.60) | 2.08 (0.62)
  Day 365 Cohort (n=41, 35) | 2.02 (0.60) | 2.08 (0.60)

3. Secondary Outcome: Adjusted Mean Change From Baseline in DAS28 CRP During Double-Blind Treatment
Description: Mean baseline DAS28 CRP values for the cohort of participants with serum samples available at that timepoint. DAS 28 is a continuous variable which is a composite of 4 variables: number of tender joints out of 28, number of swollen joints out of 28 joints, CRP in mg/L and subject assessment of disease activity measure on a VAS of 100 mm. The DAS28 provides a score on a scale from 0 to 10 indicating the current activity of the rheumatoid arthritis (>5.1=high disease activity; <3.2=low disease activity; <2.6=remission).
Time Frame: Baseline, Days 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365
Population: Number of participants analyzed=number of participants randomized; n=the number of participants with available DAS28 CRP scores at that time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
units on a scale
  Day 29 (n=45, 40) | 0.24 (0.10) | 0.06 (0.10)
  Day 57 (n=47, 37) | 0.05 (0.09) | 0.14 (0.10)
  Day 85 (n=46, 42) | 0.13 (0.10) | 0.21 (0.10)
  Day 113 (n=49, 39) | 0.02 (0.09) | 0.25 (0.10)
  Day 141 (n=47, 40) | 0.32 (0.10) | 0.29 (0.11)
  Day 169 (n=46, 36) | 0.13 (0.09) | 0.26 (0.11)
  Day 197 (n=44, 38) | 0.09 (0.09) | 0.22 (0.09)
  Day 225 (n=44, 38) | 0.25 (0.10) | 0.29 (0.10)
  Day 253 (n=46, 37) | 0.23 (0.09) | 0.14 (0.10)
  Day 281 (n=45, 38) | 0.18 (0.08) | 0.05 (0.09)
  Day 309 (n=45, 37) | 0.07 (0.08) | 0.09 (0.09)
  Day 337 (n=44, 36) | 0.26 (0.11) | 0.29 (0.13)
  Day 365 (n=41, 35) | 0.39 (0.11) | 0.16 (0.12)
Statistical Analysis 1: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 29; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted difference = 0.18, 95% CI 2-sided [-0.11 to 0.46] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 2: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 57; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.09, 95% CI 2-sided [-0.34 to 0.17] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 3: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 85; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.08, 95% CI 2-sided [-0.37 to 0.20] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 4: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 113; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.23, 95% CI 2-sided [-0.50 to 0.04] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 5: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 141; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = 0.03, 95% CI 2-sided [-0.26 to 0.32] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 6: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 169; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.13, 95% CI 2-sided [-0.41 to 0.15] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 7: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 197; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.12, 95% CI 2-sided [-0.38 to 0.13] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 8: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 225; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.04, 95% CI 2-sided [-0.32 to 0.25] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 9: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 253; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = 0.08, 95% CI 2-sided [-0.19 to 0.36] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 10: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 281; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = 0.13, 95% CI 2-sided [-0.12 to 0.38] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 11: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 309; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.03, 95% CI 2-sided [-0.27 to 0.22] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 12: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 337; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = -0.03, 95% CI 2-sided [-0.37 to 0.31] — Change from Baseline = Post-baseline - Baseline value
Statistical Analysis 13: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Day 365; Test type: Superiority or Other; ANCOVA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Adjusted Difference = 0.23, 95% CI 2-sided [-0.09 to 0.55] — Change from Baseline = Post-baseline - Baseline value

4. Secondary Outcome: Percentage of Participants With 2 Consecutive DAS 28 CRP Scores ≥ 3.2 (Loss of Low Disease Activity Status)
Description: DAS 28 is a continuous variable which is a composite of 4 variables: number of tender joints out of 28, number of swollen joints out of 28 joints, CRP in mg/L and subject assessment of disease activity measure on a VAS of 100 mm. The DAS28 provides a score on a scale from 0 to 10 indicating the current activity of the rheumatoid arthritis (>5.1=high disease activity; <3.2=low disease activity; <2.6=remission).
Time Frame: After 12 months of treatment
Population: Number of participants analyzed= number of participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants | 22.4 [11.7 to 33.1] | 22.0 [10.5 to 33.5]
Statistical Analysis 1: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Test type: Superiority or Other; normal approximation; For 95% CI: normal approximation with continuity correction; estimate of difference = 0.4, 95% CI 2-sided [-17.2 to 18.0]

5. Secondary Outcome: Percentage of Participants Given Additional DMARD Therapy During Double-Blind Treatment
Description: Additional DMARD therapy is defined as a re-introduction of methotrexate (MTX), an increase of at least 2.5 mg of MTX, or the addition of at least 1 DMARD.
Time Frame: After 12 months of treatment
Population: Number of participants analyzed= number of participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants | 3.4 [-1.2 to 8.1] | 12.0 [3.0 to 21.0]
Statistical Analysis 1: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Test type: Superiority or Other; normal approximation; For 95% CI: normal approximation with continuity correction; estimate of difference = -8.6, 95% CI 2-sided [-20.3 to 3.2]

6. Secondary Outcome: Percentage of Participants Who at Any Time During Double-Blind Treatment Were Given 2 or More Courses of High-Dose Steroids
Description: A course of high dose steroids is defined as a course of intramuscular, intravenous, or high dose oral corticosteroids (use of > 10 mg/day equivalent of prednisone for a minimum of 3 consecutive days or for those subjects who had continued use for long durations of time, each course was determined by 28 day intervals).
Time Frame: After 12 months of treatment
Population: Number of participants analyzed= number of participants randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants | 0 [0 to 0] | 0 [0 to 0]

7. Primary Outcome: Time to Disease Relapse Through Month 12 (Kaplan-Meier Cumulative Percentage of Events of Disease Relapse)
Description: An event of disease relapse was defined as additional Disease-modifying antirheumatic drug (DMARD) therapy given, or 2 or more courses of high steroids given, or return to abatacept 10 mg/kg (rescue medication given), or DAS28 C-reactive protein (CRP) score >=3.2 at 2 consecutive visits. Time to disease relapse was evaluated using life tables (Kaplan-Meier Cumulative Percentage of Events of Disease Relapse).
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: Number of participants analyzed=number of participants randomized. n=number of participants at risk at the end of a specified month.
Measure: Number; unit: Percentage of Events
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
Percentage of Events
  Month 1 (n=55, 49) | 5.17 | 2.00
  Month 2 (n=52, 47) | 8.65 | 4.00
  Month 3 (n=51, 42) | 10.41 | 12.35
  Month 4 (n=50, 38) | 12.17 | 22.78
  Month 5 (n=47, 35) | 13.96 | 26.96
  Month 6 (n=42, 33) | 23.11 | 31.13
  Month 7 (n=41, 32) | 24.94 | 33.22
  Month 8 (n=40, 31) | 26.77 | 33.22
  Month 9 (n=38, 31) | 30.43 | 33.22
  Month 10 (n=37, 31) | 32.27 | 33.22
  Month 11 (n=37, 30) | 32.27 | 35.37
  Month 12 (n=36, 28) | 32.27 | 35.37
Statistical Analysis 1: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Through Month 12; Test type: Superiority or Other; Cox proportional hazards model; Hazard Ratio (HR) = 0.870, 95% CI 2-sided [0.45 to 1.69] — Hazard ratio determined by a Cox proportional hazards model with treatment as the only covariate

8. Secondary Outcome: Percentage of Participants Given Rescue Medication Therapy During Double-Blind Treatment
Description: All subjects in the sub-study randomized to receive double-blind abatacept 5 mg/kg or 10 mg/kg. Subjects rescued to open-label treatment received abatacept 10 mg/kg.
Time Frame: After 12 months of treatment
Population: Number of participants analyzed= number of participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants | 6.9 [0.4 to 13.4] | 8.0 [0.5 to 15.5]
Statistical Analysis 1: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Test type: Superiority or Other; normal approximation; For 95% CI: normal approximation with continuity correction; estimate of difference = -1.1, 95% CI 2-sided [-12.9 to 10.7]

9. Secondary Outcome: Percentage of Participants Who Modified Therapy During Double-Blind Treatment
Description: Modified therapy=additional DMARD therapy, 2 or more courses of high dose steroids or rescue medication. Additional DMARD therapy=re-introduction of methotrexate (MTX), an increase of at least 2.5 mg of MTX, or the addition of at least 1 DMARD. A course of high dose steroids=a course of intramuscular, intravenous, or high dose oral corticosteroids (use of > 10 mg/day equivalent of prednisone for a minimum of 3 consecutive days or for those subjects who had continued use for long durations of time, each course was determined by 28 day intervals). Rescue medication=abatacept 10 mg/kg.
Time Frame: After 12 months of treatment
Population: Number of participants analyzed= number of participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants | 10.3 [2.5 to 18.2] | 18.0 [7.4 to 28.6]
Statistical Analysis 1: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Test type: Superiority or Other; normal approximation; 95% CI: normal approximation with continuity correction; estimate of difference = -7.7, 95% CI 2-sided [-22.6 to 7.3]

10. Secondary Outcome: Percentage of Participants Who Lost Remission Status
Description: Loss of remission is defined as DAS 28 CRP >=2.6.
Time Frame: After 12 months of treatment
Population: Number of participants analyzed= number of participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants | 53.4 [40.6 to 66.3] | 64.0 [50.7 to 77.3]
Statistical Analysis 1: Comparison: Abatacept (10 mg/kg) vs Abatacept (5 mg/kg); Test type: Superiority or Other; normal approximation; 95% CI: normal approximation with continuity correction; estimate of difference = -10.6, 95% CI 2-sided [-31.1 to 10.0]

11. Secondary Outcome: Steady-state Trough Serum Concentration (Cmin) of Abatacept During Double-Blind Treatment
Time Frame: Day 701 of the main study; sub-study Days 1, 85, 169, 253
Population: Number of participants analyzed= number of participants randomized; n =randomized participants with measurement at given time point. For the Day 701 measure, one apparent outlier sample was deleted..
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
ng/mL
  Main Study Day 701 (n=41, 36) | 22992.0 (9722.1) | 21713.5 (9520.5)
  Sub-Study Day 1 (n=46, 41) | 22213.0 (9275.8) | 23620.7 (9648.0)
  Sub-Study Day 85 (n=47, 43) | 24919.5 (14516.2) | 11922.1 (5681.8)
  Sub-Study Day 169 (n=48, 43) | 25725.7 (18500.5) | 9959.2 (5045.0)
  Sub-Study Day 253 (n=47, 42) | 28524.7 (19989.9) | 13516.2 (6564.6)

12. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, and Discontinuations During Double-Blind Treatment
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. Related AE/SAE=Certain, Probable, Possible, or Missing. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From start of substudy up to 56 days post last dose in the double-blind period or start of the open-label rescue period, whichever occurred first until end of study (study duration was 115 weeks)
Population: Number of participants analyzed = All treated participants during the double-blind period.
Measure: Number; unit: percentage of participants
Groups:
- Abatacept (10 mg/kg): All participants in the sub-study treated with double-blind abatacept 10 mg/kg
- Abatacept (5 mg/kg): All participants in the sub-study treated with double-blind abatacept 5 mg/kg
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants
  Deaths | 0 | 2.0
  SAEs | 5.2 | 6.0
  Related SAEs | 1.7 | 0
  Discontinued due to SAEs | 0 | 2.0
  AEs | 65.5 | 50.0
  Related AEs | 20.7 | 10.0
  Discontinued due to AEs | 0 | 2.0

13. Secondary Outcome: Percentage of Participants With Infection and Infestation AEs Reported During Double-Blind Treatment
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. Infection and Infestation AEs = any AE within the System Organ Class Infection and Infestation.
Time Frame: as for outcome 12
Population: Number of participants analyzed = All treated participants during the double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants
  Total Participants with Infection and Infestation | 37.9 | 26.0
  Upper Respiratory Tract Infection | 5.2 | 12.0
  Nasopharyngitis | 5.2 | 6.0
  Influenza | 5.2 | 4.0
  Bronchitis | 5.2 | 2.0
  Urinary Tract Infection | 3.4 | 4.0
  Onychomycosis | 3.4 | 2.0
  Pharyngitis | 3.4 | 2.0
  Rhinitis | 3.4 | 2.0
  Ear Infection | 3.4 | 0
  Vaginal Infection | 3.4 | 0
  Appendicitis | 1.7 | 0
  Furuncle | 1.7 | 0
  Pneumonia | 1.7 | 0
  Sinusitis Bacterial | 1.7 | 0
  Endocarditis | 0 | 2.0
  Fungal Skin Infection | 0 | 2.0
  Herpes Simplex | 0 | 2.0
  Labyrinthitis | 0 | 2.0
  Oral Herpes | 0 | 2.0
  Respiratory Tract Infection | 0 | 2.0
  Sinusitis | 0 | 2.0

14. Secondary Outcome: Percentage of Participants With Malignant Neoplasms Reported During Double-Blind Treatment
Description: All neoplasms were assessed by medical review as to whether or not the event was malignant.
Time Frame: as for outcome 12
Population: Number of participants analyzed = All treated participants during the double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants | 0 | 0

15. Secondary Outcome: Percentage of Participants With Prespecified Acute Infusional Adverse Events (AIAEs) During Double-Blind Treatment, by Intensity
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. Acute Infusional AE= a subset of the peri-infusional AEs with onset during the first hour after the start of the study drug infusion. A total of 105 infusional events were prespecified in the protocol.
Time Frame: as for outcome 12
Population: Number of participants analyzed = All treated participants during the double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants
  Total Participants with AIAEs (mild) | 0 | 2.0
  Total Participants with AIAEs (moderate) | 0 | 0
  Total Participants with AIAEs (severe) | 0 | 0
  Total Participants with AIAEs (very severe) | 0 | 0
  Vascular Disorders - Hypertension (mild) | 0 | 2.0
  Vascular Disorders - Hypertension (moderate) | 0 | 0
  Vascular Disorders - Hypertension (severe) | 0 | 0
  Vascular Disorders - Hypertension (very severe) | 0 | 0
  Vascular Disorders - Hypertension (unknown) | 0 | 0

16. Secondary Outcome: Percentage of Participants With Prespecified Peri-Infusional Adverse Events (PAIAEs) During Double-Blind Treatment, by Intensity
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. Peri-infusional AE=a pre-specified infusional AE occuring during the first 24 hours after the start of study drug infusion.A total of 105 infusional events were prespecified in the protocol. GDASC=General Disorders and Administration Site Conditions, RTMD=Respiratory, Thoracic and Mediastinal Disorders.
Time Frame: as for outcome 12
Population: Number of participants analyzed = All treated participants during the double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants
  Total Participants with PIAEs (mild) | 6.9 | 4.0
  Total Participants with PIAEs (moderate) | 1.7 | 0
  Total Participants with PIAEs (severe) | 0 | 0
  Total Participants with PIAEs (very severe) | 0 | 0
  Gastrointestinal Disorders, Nausea (mild) | 1.7 | 0
  Gastrointestinal Disorders, Nausea (moderate) | 0 | 0
  Gastrointestinal Disorders, Nausea (severe) | 0 | 0
  Gastrointestinal Disorders, Nausea (very severe) | 0 | 0
  Gastrointestinal Disorders, Vomiting (mild) | 1.7 | 0
  Gastrointestinal Disorders, Vomiting (moderate) | 0 | 0
  Gastrointestinal Disorders, Vomiting (severe) | 0 | 0
  Gastrointestinal Disorders, Vomiting (very severe) | 0 | 0
  Nervous System Disorders, Dizziness (mild) | 1.7 | 0
  Nervous System Disorders, Dizziness (moderate) | 0 | 0
  Nervous System Disorders, Dizziness (severe) | 0 | 0
  Nervous System Disorders, Dizziness (very severe) | 0 | 0
  Nervous System Disorders, Headache (mild) | 0 | 0
  Nervous System Disorders, Headache (moderate) | 1.7 | 0
  Nervous System Disorders, Headache (severe) | 0 | 0
  Nervous System Disorders, Headache (very severe) | 0 | 0
  GDASC, Malaise (mild) | 1.7 | 0
  GDASC, Malaise (moderate) | 0 | 0
  GDASC, Malaise (severe) | 0 | 0
  GDASC, Malaise (very severe) | 0 | 0
  GDASC, Chest Pain (mild) | 0 | 2.0
  GDASC, Chest Pain (moderate) | 0 | 0
  GDASC, Chest Pain (severe) | 0 | 0
  GDASC, Chest Pain (very severe) | 0 | 0
  RTMD, Asthma (mild) | 1.7 | 0
  RTMD, Asthma (moderate) | 0 | 0
  RTMD, Asthma (severe) | 0 | 0
  RTMD, Asthma (very severe) | 0 | 0
  RTMD, Cough (mild) | 1.7 | 0
  RTMD, Cough (moderate) | 0 | 0
  RTMD, Cough (severe) | 0 | 0
  RTMD, Cough (very severe) | 0 | 0
  Vascular Disorders, Hypertension (mild) | 0 | 2.0
  Vascular Disorders, Hypertension (moderate) | 0 | 0
  Vascular Disorders, Hypertension (severe) | 0 | 0
  Vascular Disorders, Hypertension (very severe) | 0 | 0

17. Secondary Outcome: Percentage of Participants With Pre-specified Autoimmune Disorders (ADs) Reported During Double-Blind Treatment, by Intensity
Description: A total of 127 autoimmune disorders were prespecified in the protocol. MCTD=Musculoskeletal and Connective Tissue Disorders
Time Frame: as for outcome 12
Population: Number of participants analyzed = All treated participants during the double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants
  Total Participants with ADs (mild) | 0 | 4.0
  Total Participants with ADs (moderate) | 0 | 0
  Total Participants with ADs (severe) | 0 | 0
  Total Participants with ADs (very severe) | 0 | 0
  Eye Disorders - Episcleritis (mild) | 0 | 2.0
  Eye Disorders - Episcleritis (moderate) | 0 | 0
  Eye Disorders - Episcleritis (severe) | 0 | 0
  Eye Disorders - Episcleritis (very severe) | 0 | 0
  MCTDs - Sjogren's Syndrome (mild) | 0 | 2.0
  MCTDs - Sjogren's Syndrome (moderate) | 0 | 0
  MCTDs - Sjogren's Syndrome (severe) | 0 | 0
  MCTDs - Sjogren's Syndrome (very severe) | 0 | 0

18. Secondary Outcome: Percentage of Participants With Laboratory Values Meeting the Marked Abnormality Criteria During Double-Blind Treatment
Description: Not evaluated: high hemoglobin,high hematocrit,high erythrocytes,high neutrophils+bands(N+B),low monocytes,low basophils,low eosinophils,low alkaline phosphatase(ALP),low aspartate aminotransferase(AST),low alanine aminotransferase(ALT),low G-Glutamyl transferase(GGT),low total bilirubin,low blood urea nitrogen,low creatinine,high albumin,low uric acid,low urine protein,low urine glucose,low urine blood,low urine leukocyte esterase,low urine white blood cells,low red blood cells.Pre Rx=pretreatment,(*)Lymphocytes(c/uL):Low<.750x10^3,High>7.50x10^3.(*)Eosinophils:>.750x10^3 c/uL.
Time Frame: as for outcome 12
Population: Number of participants analyzed = All treated participants during the double-blind period; n=number of participants with specific measure
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 58 | 50
percentage of participants
  Hemoglobin, Low: >3 g/dL ↓ from pre rx (n=51, 48) | 0 | 0
  Hematocrit, Low: <0.75 x pre rx (n=51, 48) | 0 | 0
  Erythrocytes, Low: <0.75 x pre rx (n=51, 48) | 0 | 0
  ALP, High: >2 x upper limit normal (ULN)(n=52, 47) | 0 | 0
  Total Calcium, Low: <0.8 x Lower LN(LLN)(n=52, 47) | 0 | 0
  Platelet Count, Low: <0.67 x LLN (n=51, 48) | 0 | 0
  Platelet Count, High: >1.5 x ULN (n=51, 48) | 0 | 0
  Leukocytes, Low: <0.75 x LLN (n=51, 48) | 0 | 0
  N+B (absolute), Low: < 1.00 x 10^3 c/uL (n=55, 49) | 0 | 0
  Lymphocytes (absolute), Low (*) (n=55, 49) | 1.8 | 2.0
  Lymphocytes (absolute), High (*) (n=55, 49) | 0 | 0
  Monocytes (absolute), High: >2000/mm^3 (n=55, 49) | 0 | 0
  Basophils (absolute), High: > 400/mm^3 (n=55, 49) | 0 | 0
  Eosinophils (absolute), High (*) (n=55, 49) | 5.5 | 2.0
  AST, High: >3 x ULN (n=52, 47) | 0 | 0
  ALT, High: >3 x ULN (n=52, 47) | 0 | 0
  GGT, High: >2 x ULN (n=52, 47) | 0 | 0
  Bilirubin Total, High: >1.5 x ULN (n=52, 46) | 0 | 0
  Blood Urea Nitrogen, High: >2 x pre rx (n=52, 47) | 0 | 0
  Serum Sodium, Low: <0.95 x LLN (n=52, 47) | 0 | 0
  Serum Sodium, High: >1.05 x ULN, (n=52, 47) | 0 | 0
  Serum Potassium, Low: <0.9 x LLN (n=52, 47) | 0 | 0
  Serum Potassium, High: >1.1 x ULN (n=52, 47) | 0 | 2.1
  Serum Chloride, Low: <0.9 x LLN (n=52, 47) | 0 | 0
  Serum Chloride, High: >1.1 x ULN, (n=52, 47) | 0 | 0
  Total Calcium, High: >1.2 x ULN (n=52, 47) | 0 | 0
  Inorganic Phosphorus, Low: <0.75 x LLN (n=52, 47) | 0 | 0
  Inorganic Phosphorus, High: >1.25 x ULN (n=52, 47) | 0 | 0
  Serum Glucose, Low: <65 mg/dL (n=55, 48) | 5.5 | 6.3
  Serum Glucose, High: >220 mg/dL (n=55, 48) | 3.6 | 4.2
  Total Protein, Low: <0.9 x LLN (n=52, 47) | 0 | 0
  Total Protein, High: >1.1 x ULN (n=52, 47) | 0 | 0
  Albumin, Low: <0.9 x LLN (n=52, 47) | 0 | 0
  Uric Acid, High: >1.5 x ULN (n=52, 47) | 0 | 0
  Urine Protein, High: >=2-4 (n=55, 47) | 1.8 | 6.4
  Urine Glucose, High: >=2-4 (n=55, 47) | 5.5 | 0
  Urine Blood, High: >=2-4 (n=55, 47) | 12.7 | 10.6
  Urine Leukocyte Esterase, High: >=2-4 (n=20, 16) | 15.0 | 25.0
  Urine White Blood Cells, High: >=2-4 (n=22, 14) | 45.5 | 14.3
  Urine Red Blood Cells, High: >=2-4 (n=22, 14) | 22.7 | 28.6

19. Secondary Outcome: Clinically Significant Changes in Vital Signs and Physical Findings
Description: Clinical significance was determined by investigator. Parameters include blood pressure, heart rate, respiration rate, and temperature.
Time Frame: as for outcome 12
Population: This analysis was not done because clinically significant changes in vital signs and physical findings were reported as adverse events.
Measure: Number; unit: participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Participants With Positive Antibody Responses to Abatacept (Electrochemiluminescence [ECL] Method) During Double-Blind Treatment
Description: A positive antibody response to Abatacept (measured by the ECL assay) is further classified as a positive response for either Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) and Possibly immunoglobulin (Ig)' or 'Ig and/or Junction Region'
Time Frame: After 12 months of treatment
Population: Number of participants analyzed= Number of participants with available immunogenicity measurements
Measure: Number; unit: participants
Arm/Group | Abatacept (10 mg/kg) | Abatacept (5 mg/kg)
Number analyzed (Participants) | 56 | 49
participants
  CTLA4 and Possibly IG | 4 | 1
  IG and/or Junction Region | 0 | 1

ADVERSE EVENTS:
Arm/Group | Abatacept 5mg/kg (ST) | Abatacept 10mg/kg (ST) | Abatacept 10mg/kg (Open-Label)
Serious Adverse Events (participants affected / at risk) | 3/50 | 3/58 | 2/8
Other Adverse Events (participants affected / at risk) | 17/50 | 18/58 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 5mg/kg (ST) (N=50) | Abatacept 10mg/kg (ST) (N=58) | Abatacept 10mg/kg (Open-Label) (N=8)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0 | 0
Acquired Claw Toe (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 5mg/kg (ST) (N=50) | Abatacept 10mg/kg (ST) (N=58) | Abatacept 10mg/kg (Open-Label) (N=8)
Conjunctivitis (Eye disorders) | 2 | 0 | 1
Xerophtalmia (Eye disorders) | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 3 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 0
Influenza (Infections and infestations) | 2 | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 3 | 0
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.